CLINICAL TRIAL: NCT01009281
Title: A 52 Week Open Label Extension Study to Evaluate the Safety and Tolerability of AIN457 (Anti IL-17 Monoclonal Antibody) in Patients With Moderate to Severe Crohn's Disease
Brief Title: An Open Label Safety and Tolerability Study of AIN457 in Patients With Moderate to Severe Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457A2202E1; EudraCT number: 2009-011621-14
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Results first posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Crohn's Disease; Inflammatory Bowel Disease
Keywords: Crohn's Disease; Crohns; Bowel disease; digestive disorders; auto immune; diarrhea; Inflammatory Bowel Disease (IBD); gastrointestinal diseases; digestive system diseases; Antibody; IL 17; anti IL-17; monoclonal antibody; Crohn's Disease (Chron's, CD)
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Intestinal Diseases; Digestive System Diseases; Diarrhea; Gastrointestinal Diseases | interventions — secukinumab

ARMS (1):
- AIN457 (Experimental)
  Interventions: Drug: AIN457

INTERVENTIONS:
Drug: AIN457

SUMMARY:
This study will assess the safety and tolerability of AIN457 in patients with moderate to severe Crohn's disease who already participated and completed the core trial CAIN457A2202.

ELIGIBILITY:
Inclusion Criteria:

* Patients who participate and complete the core CAIN457A2202 study up to and including Visit 11 (end of study), may enter the extension study upon signing informed consent.

Exclusion Criteria:

* Patients for whom continued treatment with AIN457 is not considered appropriate by the treating physician.
* Patients who were non-compliant or who demonstrated a major protocol violation in the core CAIN457A2202 study
* Patients who discontinued from the core CAIN457A2202 study before Visit 8 (day 43).

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-10-30 (Actual); Primary Completion 2010-08-19 (Actual); Study Completion 2010-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (5):
  - Conneticut Gastroenterology Institute, 39 Brewster Road, Bristol, Connecticut
  - Long Island Clinical Research Associates, LLP, Great Neck, New York
  - Mount Sinai, One Gustave L. Levy Place, Box 1118, New York, New York
  - UNC School of Medicine, Room 7200 MBRB, 103 Mason Farm Road,, Chapel Hill, North Carolina
  - Wake Research Asspcoates. ::C. 3100 Duraleigh Road, Suite 304, Raleigh, North Carolina

REFERENCES:
- [Derived] Hueber W, Sands BE, Lewitzky S, Vandemeulebroecke M, Reinisch W, Higgins PD, Wehkamp J, Feagan BG, Yao MD, Karczewski M, Karczewski J, Pezous N, Bek S, Bruin G, Mellgard B, Berger C, Londei M, Bertolino AP, Tougas G, Travis SP; Secukinumab in Crohn's Disease Study Group. Secukinumab, a human anti-IL-17A monoclonal antibody, for moderate to severe Crohn's disease: unexpected results of a randomised, double-blind placebo-controlled trial. Gut. 2012 Dec;61(12):1693-700. doi: 10.1136/gutjnl-2011-301668. Epub 2012 May 17. PMID 22595313
- See also: Related Info — http://www.NovartisClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 centers in 3 countries USA, Canada, Poland between 30-August-2009 (first participant enrolled) to 19-August-2010 (Last participant completed).
Pre-assignment Details: A total of 7 participants enrolled in the study. All seven participants were discontinued due to early termination of the core study (CAIN457A2202 [NCT00584740]) due to lack of efficacy.
Groups:
- Secukinumab: Participants received 3 milligrams per kilogram (mg/kg) of intravenous (IV) secukinumab once every 4 weeks (q4wk) up to one year of treatment.
Period: Overall Study
Arm/Group | Secukinumab
Started | 7
Completed | 0
Not Completed | 7
Not completed — Administrative problems | 7

BASELINE CHARACTERISTICS:
Population: Safety analysis set consisted of all participants who received at least one dose of study drug.
Arm/Group | Secukinumab
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.9 (15.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: From Start of the Study up to Study Termination (up to 42 Weeks)
Population: Safety analysis set consisted of all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab
Number analyzed (Participants) | 7
Participants | 3

2. Secondary Outcome: Number of Participants With Anti-AIN457 Antibodies
Description: Anti-AIN457 antibodies were assessed in serum.
Time Frame: From Start of the Study up to Study Termination (up to 42 Weeks)
Population: Safety analysis set consisted of all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab
Number analyzed (Participants) | 7
Participants | NA — Due to significant delays in sample processing this analysis was not conducted, hence results are not available.

3. Secondary Outcome: Change From Baseline in Concentration of Interleukin 17 (IL-17)
Time Frame: Baseline up to Study Termination (up to 42 Weeks)
Population: Safety analysis set consisted of all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab
Number analyzed (Participants) | 7
Participants | NA — Due to technical issues this analysis could not be conducted and therefore no results are available for inclusion in this report.

4. Secondary Outcome: Change From Baseline in Levels of Fecal Calprotectin and Lactoferrin
Time Frame: Baseline up to Study Termination (up to 42 Weeks)
Population: Safety analysis set consisted of all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab
Number analyzed (Participants) | 7
Participants | NA — Results are unavailable as the analysis could not be performed due to early termination and the small number of participants in the study

5. Secondary Outcome: Change From Baseline in C-Reactive Protein Levels
Time Frame: Baseline up to Study Termination (up to 42 Weeks)
Population: Safety analysis set consisted of all participants who received at least one dose of study drug. Here, the number of participants analyzed refer to the participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | Secukinumab
Number analyzed (Participants) | 6
milligram per liter (mg/L) | 14.2 (20.54)

6. Secondary Outcome: Maximum (Peak) Observed Steady-State Drug Concentration in the Plasma, Blood, Serum, or Other Body Fluids During Multiple Dosing [Amount x Volume-1] (Cmax,ss)
Time Frame: Pre-dose, post dose on week 44 (end of infusion)
Population: Pharmacokinetic data analysis included all participants with evaluable pharmacokinetic data. Due to the early discontinuation of all participants, the full dataset of concentration measurements could not be obtained, analyzed and reported.
Arm/Group | Secukinumab
Number analyzed (Participants) | 0

7. Secondary Outcome: Minimum Observed Steady-State Drug Concentration in the Plasma, Blood, Serum, or Other Body Fluids at the End of the Dosing Intervals During Multiple Dosing [Amount x Volume-1] (Cmin,ss)
Time Frame: Pre-dose, post dose on week 44 (end of infusion)
Population: as for outcome 6
Arm/Group | Secukinumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From Start of the Study up to Study Termination (up to 42 weeks)
Arm/Group | Secukinumab
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab (N=7)
Abdominal distension (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Influenza like illness (General disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Depression (Psychiatric disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early as participants were discontinued prematurely due to early termination of the core trial (CAIN457A2202 [NCT00584740]). This decision was based on fulfillment of the futility criterion for lack of efficacy, assessed during a scheduled interim analysis in the core trial. Therefore, only very limited information is available from this extension study (CAIN457A2202E1 [NCT01009281]).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No